CLINICAL TRIAL: NCT00006154
Title: Randomized, Controlled, Open Label, Multi-Center Phase III Trial Comparing the Safety and Antiviral Activity of a Protease-Containing Regimen (d4T/ddI/IDV/RTV) Versus a Protease-Sparing Regimen (d4T/ddI/EFV) and the Ability of Interleukin-2 to Purge HIV From Latent Stores in Patients With Acute/Early HIV Infection
Brief Title: A Study to Evaluate the Use of a Protease Inhibitor and of Interleukin-2 (IL-2) in the Treatment of Early HIV Infection
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AI-07-001; CTN #124; 11530 (Registry Identifier: DAIDS-ES)
Record Dates: First submitted 2000-08-07; First posted 2001-08-31 (Estimated); Last update posted 2013-09-06 (Estimated); Status verified 2013-09

CONDITIONS: HIV Infections
Keywords: Interleukin-2; Didanosine; Drug Therapy, Combination; Stavudine; HIV Protease Inhibitors; Ritonavir; Indinavir; Virus Latency; Reverse Transcriptase Inhibitors; Anti-HIV Agents; abacavir; efavirenz; Acute Infection
MeSH Terms: conditions — HIV Infections | interventions — Indinavir; Ritonavir; abacavir; efavirenz; Stavudine; Didanosine; aldesleukin; Interleukin-2

ARMS (2):
- A (Experimental): Patients will receive combination antiretroviral therapy with a protease inhibitor
  Interventions: Drug: Indinavir sulfate; Drug: Ritonavir; Drug: Abacavir sulfate; Drug: Didanosine; Drug: Aldesleukin
- B (Active Comparator): Patients will receive combination antiretroviral therapy without a protease inhibitor
  Interventions: Drug: Abacavir sulfate; Drug: Efavirenz; Drug: Stavudine; Drug: Didanosine; Drug: Aldesleukin

INTERVENTIONS:
Drug: Indinavir sulfate — 400 mg tablets equaling 1600 mg daily
  Other Names: IDV
  Arms: A
Drug: Ritonavir — 100 mg liquid capsules equaling 400 mg daily
  Other Names: RTV
  Arms: A
Drug: Abacavir sulfate — 300 mg capsules equaling 600 mg daily. Administration based on individual results after 16 weeks.
  Other Names: ABC
Drug: Efavirenz — 200 mg capsules equaling 600 mg daily
  Other Names: DMP
  Arms: B
Drug: Stavudine — 30-40 mg capsules equaling 60 or 80 mg daily
  Other Names: d4T
  Arms: B
Drug: Didanosine — 250-400 mg E.coated tablets equaling 250 or 400 mg daily
  Other Names: ddI
Drug: Aldesleukin — Subcutaneous injection equaling 15 x 10^6 IU daily dose. Administration based on individual results after 16 weeks and randomization.
  Other Names: Proleukin; IL-2

SUMMARY:
The purpose of this study is to look at the effectiveness of combination anti-HIV drug therapy (with protease inhibitors [PIs] or without) in patients with early HIV infections. This study also looks at whether a drug called interleukin-2 (IL-2) can boost the immune system of these patients.

Doctors are not sure which anti-HIV drug combination is best to use in patients who have early HIV infection and have never received anti-HIV treatment. PIs are anti-HIV drugs that decrease viral load (level of HIV in the blood). However, PIs can cause serious side effects in some patients. Doctors would like to know if a drug combination that does not contain a PI is just as good as one that contains PIs.

DETAILED DESCRIPTION:
Studies have suggested that an antiretroviral drug regimen of the non-nucleoside agent efavirenz (EFV) in combination with two nucleoside analogues is effective at achieving maximal viral suppression. This provides an alternative treatment to that of the more toxic PI-containing regimen. This trial examines whether a nonPI regimen with EFV is more beneficial than a PI-containing regimen when each is used in combination with the same two nucleoside analogues. A second part of the study looks at whether the addition of IL-2 may offer immunologic benefits as a co-administered drug.

Patients are randomized to initiate antiretroviral therapy of a PI-based (stavudine/didanosine/ritonavir [RTV]/indinavir [IDV]) or nonPI-based (stavudine/didanosine/EFV) regimen. Within these treatment arms, they are stratified according to a positive or negative p24 antigen result. At Week 16, patients not achieving maximal viral suppression (lower than 50 copies/ml) have the option to add abacavir (ABC) or other drugs as intensification therapy. Those achieving virologic suppression (less than 50 copies/ml) are randomized either to receive IL-2 or not. At study entry, and after 12 months, tissue samples of CSF, lymph node, and genital secretions are obtained, with permission. Patients have physical exams, women of child-bearing potential have pregnancy tests, and blood samples are drawn at clinic visits 12-16 times a year over 3 years so that virologic and immunologic evaluations may be performed. Compensation for time and transportation is given.

ELIGIBILITY:
Inclusion Criteria

Patients may be eligible for this study if they:

* Have been infected recently with HIV. This will be determined by certain lab tests.
* Are 18 years of age or older.
* Are able to swallow a large number of pills.
* Are willing to use barrier methods of birth control (such as condoms) during the study.

Exclusion Criteria

Patients will not be eligible for this study if they:

* Abuse drugs or alcohol.
* Have any condition that, in the opinion of the investigator, could impair their ability to participate in the study.
* Are breast-feeding or pregnant.
* Have received any prior anti-HIV drugs. (However, use of anti-HIV drugs to try to prevent infection more than 6 months prior to study entry is allowed.)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 165 (Estimated)

PRIMARY OUTCOMES:
Virologic: A. Plasma viral load B. Tissue viral load (CNS, lymphoid tissues, genital tract) C. HIV DNA (proviral) levels in circulating mononuclear cells D. Phenotypic and genotypic antiretroviral drug resistance | Throughout study
Immunologic: A. Evaluation of CD4, CD8, CD45RA, CD45RO phenotypes and defined activation markers B. Evaluation of the diversity and persistence of the T cell repertoire (CD4+, CD8+) in the circulation and lymphoid tissues | Throughout study
Immunologic: C. Functional CD4+ cellular assays (class II MHC tetramers) D. Thymic regeneration as studied by the exclusion circle assay E. Evolution of Western blot banding patterns F. Evolution of anti-HIV neutralizing antibody levels | Throughout study
Clinical: A. Minor opportunistic infections or AIDS-defining conditions B. Death C. Clinical or laboratory adverse events D. Evaluation of adherence to therapy E. Evaluation of lipodystrophy | Throughout study

CONTACTS AND LOCATIONS:
Overall Officials: Rafick-Pierre Sekaly, Principal Investigator; Brian Conway, Principal Investigator
Locations (4):
- Canada (4):
  - Viridae Clinical Sciences / University of British Columbia, Vancouver, British Columbia
  - Centre de traitment d'immunodeficience, Montreal, Quebec
  - Centre Hospitalier de la Universite de Montreal (CHUM), Montreal, Quebec
  - Institut Thoracique de Montreal, Montreal, Quebec